CLINICAL TRIAL: NCT04149119
Title: Attractive Targeted Sugar Bait Phase III Trial in Mali
Brief Title: Attractive Targeted Sugar Bait Trial in Mali
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University Clinical Research Center, Mali (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Prevention
Other Study IDs: 6719882
Record Dates: First submitted 2019-10-01; First posted 2019-11-04 (Actual); Last update posted 2021-07-07 (Actual); Status verified 2021-03

CONDITIONS: Vector Transmission
Keywords: Malaria; Vector control; ATSB; Transmission; Mali
MeSH Terms: conditions — Malaria

STUDY DESIGN:
Intervention Model Description: An open-label two-arm cluster randomized controlled trial (CRCT) design will be used comparing ATSB + LLINS vs LLINS alone (standard of care). A cluster trial design is indicated given the intended community-level effect of ATSBs on malaria transmission. Universal LLIN coverage will be ensured in both arms prior to start of the study and will serve as the standard of care. Arm 1 will receive ATSBs for two years. Arm 2 will receive the standard of care of universal LLIN coverage.
  The incidence cohorts will be powered to detect a 30% reduction in incidence assuming follow-up over a two year period (see sample size section). Prevalence of infection will be powered to detect a 30% lower prevalence in the treatment arm of of the trial during each of the two post randomisation cross sectional surveys.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention arm (Experimental): ATSB+LLINs+Standard Care for Malaria case management
  Interventions: Device: Attractive Target Sugar Baits (ATSB)
- Standard arm or arm 2 (No Intervention): LLINs+Standard Care for MalarIA case management

INTERVENTIONS:
Device: Attractive Target Sugar Baits (ATSB) — Within the intervention area, a total of four ATSB station will be deployed (external wall). ATSB stations will be monitored by community health workers through weekly visit and all stations will be replaced 6months after deployment.
  Arms: Intervention arm

SUMMARY:
Globally, the female mosquitoes to be effective at transmitting malaria parasites, must have a number of characteristics including: abundance, longevity (individual mosquitoes must survive long enough after feeding on infected blood to allow the parasite time to develop and travel to the mosquito's salivary glands), capacity (each female mosquito must be both susceptible to infection with Plasmodium and able to carry enough malaria parasites in the salivary glands), contact with humans (frequently feed on humans).

Vectors in SSA are often anthropophagic and anthropophilic, and exhibit indoor biting and indoor resting behavior. Highly effective interventions against vectors have been developed and implemented at scale (e.g., indoor Residual Spraying of Insecticides [IRS] and Long Lasting Insecticide-treated Nets [LLINs]). While these interventions have contributed importantly to the reduction of malaria transmission and disease (68% and 11% respectively), none of them target outdoor-biting g and outdoor-resting mosquitoes. Given the increase in resistance to current generation of insecticides and the behavioral plasticity of vectors that results in continued malaria transmission despite high coverage of LLINs or IRS, there is a need for interventions that can supplement and complement LLINs and IRS by killing mosquitoes outside houses using other biologic mechanisms (e.g., targeting sugar feeding behavior). Finally, insecticides with novel modes of action that may be capable of restoring sensitivity to pyrethroids by killing both pyrethroid resistant and sensitive mosquitoes are required. Attractive Target Sugar Baits (ATSBs) that kill mosquitoes through the ingestion of the toxicant dinotefuran (and possibly by other ingestion toxicants that are effective when ingested) potentially fill the need for outdoor interventions with novel killing effects. This study aims to establish the efficacy and contribution of the ATSBs for controlling malaria transmission where An. gambiae s.l. and An. Funestus are the major vectors for malaria.

DETAILED DESCRIPTION:
The current dominant malaria vector control tools remain critically important and have saved many lives. Yet, they are not well-suited for malaria vectors that avoid contact with indoor insecticides by predominantly biting outdoors, by frequently biting animals, and by resting outdoors or remaining within houses only briefly when they do enter. These behaviors allow residual populations of vector mosquitoes to survive, expand, and to increasingly contribute to malaria transmission, despite high coverage. These vectors can sustain endemic transmission even if they rarely bite humans. An. arabiensis is a particularly important source of persistent residual transmission despite Long Lasting Insecticide-treated Net (LLIN) scale-up; this mosquito prefers to feed on animals, and, often bites and rests outside, and has limited indoor exposure. There is need for new vector control tools to target residual outdoor transmission.

In addition to the biological need for female Anopheles species to take a blood meal to obtain protein necessary for egg production, all Anopheles must feed regularly and frequently on liquid and carbohydrates (sugars) to survive. Common sources of liquid and sugar meals include plant tissue and floral nectar. Mosquitoes are guided to sugar sources by chemical attractants. The Attractive Target Sugar Baits (ATSBs) is designed specifically to attract the mosquito with a source of liquid and sugar and include an ingestion toxicant to then kill the mosquito. Using sugar sources to attract mosquitoes to an ingestion toxicant is a relatively simple and inexpensive, strategy that has been shown to be highly efficacious for mosquito control in a limited number of trials. Limited data suggest efficacy, even in sugar-rich environments, due to the high frequency of sugar feeding.

Early studies examined the effect of spraying ingestion toxicants on attractive flowers to use their scent as bait. While these flowers effectively attract the target mosquitoes, the impact on non-target insects, especially pollinators, can be devastating. Furthermore, this approach is not suitable where there is a lack of flowering vegetation. Subsequent studies evaluated locally available plants and fruits as attractants. While such attractants can be sprayed onto non-flowering green vegetation, further studies evaluated products (bait stations) that could be used across a wide variety of settings including indoors and in areas without suitable vegetation.

Westham Compagny recently developed a bait station that contains a plant-based mosquito attractant, sugar as a feeding stimulant, and an active ingredient (the neonicotinoid, dinotefuran) to kill the foraging vectors. The bait station has a protective membrane that covers and protects the bait from rain and dust, but that allows mosquitoes to feed through it. The Westham ATSB can remain effective in the field for at least six months and has a shelf life of greater than three years with no specific requirements for storage. This Attractive Target Sugar Bait (ATSB) is now being produced at an industrial scale, uses simple and widely available ingredients, and is environmentally friendly. The bait station was designed to have the lowest practicable material content with a high proportion of the mass being fully biodegradable. The protective membrane allows mosquitoes to feed, but it serves as a barrier to pollinators. Field studies to-date have also shown that the ATSB has a minimal impact on non-target organisms. This includes evidence specifically for the toxicant that will be used, dinotefuran. Initial environmental assessment and subsequent field trials in Mali have demonstrated that when deployed within the ATSB, the toxicant does not pose safety risks to non-target organisms, including pollinators and humans.

ATSBs may be a particularly important vector control tool in the context of insecticide resistance. Insecticide resistance for the six insecticide classes currently used in LLINs and IRS threatens malaria prevention efforts. Resistance to pyrethroids (used in LLINs and IRS) is commonly reported. If pyrethroids lose most of their efficacy, more than 55% of the benefits of vector control could be lost. ATSBs can help mitigate insecticide resistance to these contact insecticides because they can use ingestion toxicants from very different chemical classes. There are many existing ingestion toxicants that may be used in a bait station, which could facilitate resistance prevention strategies, such as rotation or combination approaches.

ELIGIBILITY:
Inclusion criteria

* . Household resident of the selected villages
* Aged 5 to 14 years of age at the time of enrollment
* All parents or guardians provide consent for their child's participant (5-14 years old)
* If age 12 - 14 years, the child also provides assent for participation
* Absence of pregnancy

Exclusion criteria

* Not resident of any household within the selected villages
* Children below 5 years old
* Aged 15 years and older
* Pregnancy
* Do not consent or assent (14 years old)

Ages: 5 Years to 14 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 2100 (Estimated)
Dates: Start 2022-05-01 (Estimated); Primary Completion 2023-12-31 (Estimated); Study Completion 2024-06-30 (Estimated)

PRIMARY OUTCOMES:
Malaria incidence per person times | Through study completion (average 2 years
  Malaria case incidence (the total number of incident malaria cases detected by RDT divided by the total person-time followed up in cohorts) will be assessed among people aged 5 to < 15 years old

SECONDARY OUTCOMES:
Incidence of malaria per person times using molecular analysis tools | Through study completion (average 2 years
  PCR will be use to assess Incidence of malaria infection among cohort participants aged 5 to <15 years.
  2. Prevalence of malaria infection among a cross sectional sample 3. Incidence rate of passively reported clinical malaria among participants of all ages, defined as the number of malaria confirmed cases (by RDT or microscopy) per 1,000 population per year, 4. Vector age structure: survivorship will be monitored by ovarian dissection to examine ovarian dilatations.
  5. Vector densities, Sporozoite rate by CS ELISA, Entomological inoculation rates (EIR), Biting profiles, Vector species composition.
  6. Durability of the ATSB stations: 1) the effectiveness of the attractant; and 2) the effective toxicity of the ATSB.
  7. Resistance to the ATSB toxicant: susceptibility to the ingestion toxicant (dinotefuran) will be evaluated on an annual basis.
  a. Insecticide resistance: Physiological resistance phenotypes, Intensity of resistance, Behavioral resistance

OTHER OUTCOMES:
Community acceptance of ATSBs in intervention area | Through study completion (average 2 years
  Removal, alteration of ATSBs stations after deployement will be assessed and reported as acceptance in terms of proportion among intervention sites during the study period (2 years)

CONTACTS AND LOCATIONS:
Overall Officials: Seydou Doumbia, PhD, Study Director — University Clinical Research Center - USTTB - Mali
Locations (1):
- University Clinical Research Center, Bamako, Mali

IPD SHARING:
Plan to Share IPD: No
The sections below provide details of data management for individual study components. All data will be stored on a secure drive in Mali and shared with PATH. All investigators and the sponsor, Inovated Vector Control Consortium (IVCC), will have access to the data. At London School of Hygien and Tropical Medicine (LSHTM), data will be retained for a minimum of 10 years following project completion as mandated by the LSHTM's policies. Data documentation and the labelled dataset will be deposited in the LSHTM data repository (http://datacompass.lshtm.ac.uk/ ) for long-term curation and preservation at the end of the project.

REFERENCES:
- [Background] Sinka ME, Bangs MJ, Manguin S, Rubio-Palis Y, Chareonviriyaphap T, Coetzee M, Mbogo CM, Hemingway J, Patil AP, Temperley WH, Gething PW, Kabaria CW, Burkot TR, Harbach RE, Hay SI. A global map of dominant malaria vectors. Parasit Vectors. 2012 Apr 4;5:69. doi: 10.1186/1756-3305-5-69. PMID 22475528
- [Background] Bhatt S, Weiss DJ, Cameron E, Bisanzio D, Mappin B, Dalrymple U, Battle K, Moyes CL, Henry A, Eckhoff PA, Wenger EA, Briet O, Penny MA, Smith TA, Bennett A, Yukich J, Eisele TP, Griffin JT, Fergus CA, Lynch M, Lindgren F, Cohen JM, Murray CLJ, Smith DL, Hay SI, Cibulskis RE, Gething PW. The effect of malaria control on Plasmodium falciparum in Africa between 2000 and 2015. Nature. 2015 Oct 8;526(7572):207-211. doi: 10.1038/nature15535. Epub 2015 Sep 16. PMID 26375008
- [Background] Ranson H, Lissenden N. Insecticide Resistance in African Anopheles Mosquitoes: A Worsening Situation that Needs Urgent Action to Maintain Malaria Control. Trends Parasitol. 2016 Mar;32(3):187-196. doi: 10.1016/j.pt.2015.11.010. Epub 2016 Jan 27. PMID 26826784
- [Background] Amek N, Bayoh N, Hamel M, Lindblade KA, Gimnig JE, Odhiambo F, Laserson KF, Slutsker L, Smith T, Vounatsou P. Spatial and temporal dynamics of malaria transmission in rural Western Kenya. Parasit Vectors. 2012 Apr 28;5:86. doi: 10.1186/1756-3305-5-86. PMID 22541138
- [Background] Moiroux N, Damien GB, Egrot M, Djenontin A, Chandre F, Corbel V, Killeen GF, Pennetier C. Human exposure to early morning Anopheles funestus biting behavior and personal protection provided by long-lasting insecticidal nets. PLoS One. 2014 Aug 12;9(8):e104967. doi: 10.1371/journal.pone.0104967. eCollection 2014. PMID 25115830
- [Background] Sougoufara S, Diedhiou SM, Doucoure S, Diagne N, Sembene PM, Harry M, Trape JF, Sokhna C, Ndiath MO. Biting by Anopheles funestus in broad daylight after use of long-lasting insecticidal nets: a new challenge to malaria elimination. Malar J. 2014 Mar 28;13:125. doi: 10.1186/1475-2875-13-125. PMID 24678587
- [Background] Huho B, Briet O, Seyoum A, Sikaala C, Bayoh N, Gimnig J, Okumu F, Diallo D, Abdulla S, Smith T, Killeen G. Consistently high estimates for the proportion of human exposure to malaria vector populations occurring indoors in rural Africa. Int J Epidemiol. 2013 Feb;42(1):235-47. doi: 10.1093/ije/dys214. Epub 2013 Feb 9. PMID 23396849
- [Background] Killeen GF. Characterizing, controlling and eliminating residual malaria transmission. Malar J. 2014 Aug 23;13:330. doi: 10.1186/1475-2875-13-330. PMID 25149656
- [Background] Killeen GF, Marshall JM, Kiware SS, South AB, Tusting LS, Chaki PP, Govella NJ. Measuring, manipulating and exploiting behaviours of adult mosquitoes to optimise malaria vector control impact. BMJ Glob Health. 2017 Apr 26;2(2):e000212. doi: 10.1136/bmjgh-2016-000212. eCollection 2017. PMID 28589023
- [Background] Zhu L, Muller GC, Marshall JM, Arheart KL, Qualls WA, Hlaing WM, Schlein Y, Traore SF, Doumbia S, Beier JC. Is outdoor vector control needed for malaria elimination? An individual-based modelling study. Malar J. 2017 Jul 3;16(1):266. doi: 10.1186/s12936-017-1920-y. PMID 28673298
- [Background] Muller GC and Galili A. (2016). Attractive toxic sugar baits (ATSB): from basic science to product- a new paradigm for vector control. Roll Back Malaria, Vector Control Working Group meeting presentation.
- [Background] Beier JC, Muller GC, Gu W, Arheart KL, Schlein Y. Attractive toxic sugar bait (ATSB) methods decimate populations of Anopheles malaria vectors in arid environments regardless of the local availability of favoured sugar-source blossoms. Malar J. 2012 Feb 1;11:31. doi: 10.1186/1475-2875-11-31. PMID 22297155
- [Background] Muller GC, Beier JC, Traore SF, Toure MB, Traore MM, Bah S, Doumbia S, Schlein Y. Field experiments of Anopheles gambiae attraction to local fruits/seedpods and flowering plants in Mali to optimize strategies for malaria vector control in Africa using attractive toxic sugar bait methods. Malar J. 2010 Sep 20;9:262. doi: 10.1186/1475-2875-9-262. PMID 20854666
- [Background] Mnzava AP, Knox TB, Temu EA, Trett A, Fornadel C, Hemingway J, Renshaw M. Implementation of the global plan for insecticide resistance management in malaria vectors: progress, challenges and the way forward. Malar J. 2015 Apr 23;14:173. doi: 10.1186/s12936-015-0693-4. PMID 25899397
- [Background] Marshall JM, White MT, Ghani AC, Schlein Y, Muller GC, Beier JC. Quantifying the mosquito's sweet tooth: modelling the effectiveness of attractive toxic sugar baits (ATSB) for malaria vector control. Malar J. 2013 Aug 23;12:291. doi: 10.1186/1475-2875-12-291. PMID 23968494
- [Background] WHO. (2017). Malaria vector control policy recommendations and their applicability to product evaluation. Geneva: WHO.
- [Background] Midega JT, Mbogo CM, Mwnambi H, Wilson MD, Ojwang G, Mwangangi JM, Nzovu JG, Githure JI, Yan G, Beier JC. Estimating dispersal and survival of Anopheles gambiae and Anopheles funestus along the Kenyan coast by using mark-release-recapture methods. J Med Entomol. 2007 Nov;44(6):923-9. doi: 10.1603/0022-2585(2007)44[923:edasoa]2.0.co;2. PMID 18047189
- [Background] Gimnig JE, Walker ED, Otieno P, Kosgei J, Olang G, Ombok M, Williamson J, Marwanga D, Abong'o D, Desai M, Kariuki S, Hamel MJ, Lobo NF, Vulule J, Bayoh MN. Incidence of malaria among mosquito collectors conducting human landing catches in western Kenya. Am J Trop Med Hyg. 2013 Feb;88(2):301-8. doi: 10.4269/ajtmh.2012.12-0209. Epub 2012 Dec 18. PMID 23249685
- [Derived] Sarrassat S, Toure M, Diarra A, Keita M, Coulibaly H, Arou AZ, Traore M, Tangara CO, Bradley J, Muller G, Majambere S, Beier JC, Vontas J, Traore SF, Diop S, Kleinschmidt I, Doumbia S. Evaluation of Attractive Targeted Sugar Baits, a new outdoor vector control strategy against malaria: Results from a cluster randomised open-label parallel arm controlled trial in Southwestern Mali. J Infect. 2025 Jul;91(1):106524. doi: 10.1016/j.jinf.2025.106524. Epub 2025 Jun 5. PMID 40482859
- [Derived] Attractive Targeted Sugar Bait Phase III Trial Group. Attractive targeted sugar bait phase III trials in Kenya, Mali, and Zambia. Trials. 2022 Aug 9;23(1):640. doi: 10.1186/s13063-022-06555-8. PMID 35945599